CLINICAL TRIAL: NCT02950532
Title: Posterior Ligament Complex Assessment Without Magnetic Resonance Image in Thoracolumbar Fractures (T11-L2): A Diagnostic Test Study to Analyze Sensitivity and Specificity
Brief Title: Posterior Ligament Complex Assessment Without Magnetic Resonance Image in Thoracolumbar Fractures
Acronym: PAM
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: AOCID_PAM
Record Dates: First submitted 2016-10-18; First posted 2016-11-01 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Spinal Deformity; Spinal Fractures; Spinal Injuries; Kyphosis
Keywords: Posterior ligamentous complex; Thoracolumbar fractures; Interspinous distance; Local kyphosis
MeSH Terms: conditions — Spinal Fractures; Spinal Injuries; Kyphosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Retrospective radiological evaluation in cases presenting A3 or A4 TL burst fractures (AOSpine classification) between T11 to L2 with or without suspected PLC injury
  Interventions: Other: Retrospective radiological evaluation

INTERVENTIONS:
Other: Retrospective radiological evaluation — Radiological evaluation will be performed in already existing imaging exams. Superior-inferior end plate angle (SIEA), vertebral body height (BH), local kyphosis (LK), inter-spinous distance (ISD) and inter-pedicular distance (IPD) will be measured in CT scans and radiographs (if available). PLC injury will be determinated with the gold standard method (MRI).

SUMMARY:
The objective of this investigation is to confirm the results obtained in a pilot study showing that certain radiological parameters based on computed tomography (CT) scans seem to reliably detect posterior ligament complex (PLC) injury without the need for Magnetic Resonance Imaging (MRI)

DETAILED DESCRIPTION:
Integrity of posterior ligament complex (PLC) has an important bearing on the treatment strategies for thoracolumbar (TL) fractures. Magnetic Resonance Imaging (MRI) is the gold standard to confirm PLC injury. The routine use of MRI has its limitations especially since in most trauma centers MRI is not the primary assessment for TL fractures due to reduced availability, increased cost and its adverse applicability in trauma setting and in case of a polytrauma. In contrast computed tomography (CT) scans are an integral part of trauma evaluation protocols, are accurate in spine fracture diagnosis and are performed in less time, making them suitable to assess polytrauma scenarios. In a recent pilot study, a number of radiological parameters based on CT scans have shown to reliably detect PLC injury when compared to MRI. The aim of the study is to reconfirm and validate these CT based parameters to assess PLC injury compared to MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years
* A3/A4 TL fracture between T11-L2 with or without PLC injury
* Pre-treatment CT scan and MRI. Radiographs (if available)
* Signed Informed consent, if required by EC/IRB

Exclusion Criteria:

* Pathological fractures
* Multilevel contiguous and non-contiguous injuries
* Fractures with obvious spinous process split indicating tension band failure such as AO type B1 injuries
* Fractures with translation injuries or dislocations such as AO type C injuries

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The participating study sites will retrospectively identify all eligible patients in the medical charts (i.e. who meet all of the inclusion and none of the exclusion criteria). If required by local regulations, patients choosing to participate will sign and date an informed consent form (ICF).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Local kyphosis (LK) and/or Inter-spinous distanceI (SD) | CT scans, MRI and x-rays were taken on admission into hospital after the patient got a thoracolumbar fracture. These images will be retrospectively analyzed (eligible images are from the date of the fracture up to 3 days after the event).
  Sensitivity of LK and/or ISD Is defined as the proportion of patients with PLC injury correctly diagnosed by an increase in LK and/or ISD difference compared to MRI. The Specificity si defined as the proportion of patients with PLC injury correctly diagnosed by an increase in LK and/or ISD difference compared to MRI. The gold standard is a diagnostic test and it is the best accepted test that is assumed to be able to determine the true disease state. It is considered as the reference method or the best test available.

SECONDARY OUTCOMES:
Sensitivity and specificity of superior-inferior end plate angle (SIEA) | CT scans, MRI and x-rays were taken on admission into hospital after the patient got a thoracolumbar fracture. These images will be retrospectively analyzed (eligible images are from the date of the fracture up to 3 days after the event).
  Is defined as the proportion of patients with PLC injury correctly diagnosed by a increase in SIEA compared to MRI.
Sensitivity and specificity of vertebral body height (BH) | CT scans, MRI and x-rays were taken on admission into hospital after the patient got a thoracolumbar fracture. These images will be retrospectively analyzed (eligible images are from the date of the fracture up to 3 days after the event).
  Is defined as the proportion of patients with PLC injury correctly diagnosed by an decrease in BH compared to MRI.
Sensitivity and specificity of inter-pedicular distance (IPD) | CT scans, MRI and x-rays were taken on admission into hospital after the patient got a thoracolumbar fracture. These images will be retrospectively analyzed (eligible images are from the date of the fracture up to 3 days after the event).
  Is defined as the proportion of patients with PLC injury correctly diagnosed by a increase in IPD compared to MRI.

OTHER OUTCOMES:
Accuracy of CT scan measurements | CT scans, MRI and x-rays were taken on admission into hospital after the patient got a thoracolumbar fracture. These images will be retrospectively analyzed (eligible images are from the date of the fracture up to 3 days after the event).
  Accuracy describes how closely the measured value is to the true value and is an indicator of systematic errors. The accuracy of measurements of each CT scan parameter will be compared between the participating sites.
Inter-rater reliability | CT scans, MRI and x-rays were taken on admission into hospital after the patient got a thoracolumbar fracture. These images will be retrospectively analyzed (eligible images are from the date of the fracture up to 3 days after the event).
  The inter-rater reliability is defined as the percent agreement between the measurements of the different parameters by the different observers. The CT scans and radiographs (if available) distributed to the participating sites will be measured at each site by all participating MDs within each team or at least by one trained PI.

CONTACTS AND LOCATIONS:
Overall Officials: Shanmuganathan Rajasekaran, Prof. MD, Principal Investigator — Ganga Hospital; Test Testing, MD, Study Chair — TESTING
Locations (5):
- The 1st Affiliated Hospital of Zhejiang University, Hangzhou, China
- Assiut Universtiy Hospitals, Asyut, Egypt
- Ganga Hospital, Coimbatore, India
- Uijeongbu St. Mary's Hospital, Uijeongbu-si, South Korea
- Royal Victoria Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Publication